CLINICAL TRIAL: NCT06217380
Title: Feasibility and Acceptability of Oxygen Saturation Monitoring Using Masimo SafetyNet Alert (MSNA) in a Supportive Housing Program
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor's Decision
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: SAFE0004
Record Dates: First submitted 2023-11-14; First posted 2024-01-22 (Actual); Results first posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-07

CONDITIONS: Opioid Use

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Masimo SafetyNet Alert (MSNA) (Experimental): All subjects who are enrolled into the test group (excluding staff participants) and participate in data collection receive the noninvasive Masimo SafetyNet Alert (MSNA)
  Interventions: Device: Masimo SafetyNet Alert (MSNA)

INTERVENTIONS:
Device: Masimo SafetyNet Alert (MSNA) — This study will explore the feasibility of implementing the Masimo SafetyNet Alert (MSNA) oxygen saturation monitoring system and the acceptance of MSNA by individuals living in a supportive housing program, who inject opioids.

SUMMARY:
This Clinical Trial will evaluate the Feasibility and Acceptability of Oxygen Saturation Monitoring using Masimo SafetyNet Alert (MSNA) in a Supportive Housing Program

ELIGIBILITY:
Inclusion Criteria for Client Participants:

* Participants who are18 years of age or greater
* Participants housed within a supportive housing program who intend to inject opioids
* Participants who have given verbal informed consent to participate in the study

Inclusion Criteria for Staff Participants:

* Participant is research staff and/or Rita Thompson Residence staff
* Participant is willing to give implied consent by reading and completing the staff survey

Exclusion Criteria for Client Participants:

* Participants deemed not suitable for the study at the discretion of the principal investigator, research staff or housing program nurses/staff
* Participants with skin abnormalities at the planned application sites that may interfere with sensor application, per directions-for-use (DFU) or trans-illumination of the site, such as psoriasis, eczema, angioma, burns, scar tissue, substantial skin breakdown, nail polish, acrylic nails, infections, or other abnormalities that may interfere with MSNA functioning
* Participants with known allergic reactions to foam/rubber products and/or adhesive tape

Exclusion Criteria for Staff Participants:

-None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Vanier, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: No staff participants were enrolled in this study prior to termination.
Groups:
- Masimo SafetyNet Alert (MSNA): All subjects who are enrolled into the test group and participate in data collection receive the noninvasive Masimo SafetyNet Alert (MSNA)
  Masimo SafetyNet Alert (MSNA): This study will explore the feasibility of implementing the Masimo SafetyNet Alert (MSNA) oxygen saturation monitoring system and the acceptance of MSNA by individuals living in a supportive housing program, who inject opioids.
Period: Overall Study
Arm/Group | Masimo SafetyNet Alert (MSNA)
Started | 10
Completed | 6
Not Completed | 4
Not completed — Death: Unrelated to the device. The subject was enrolled but did not start any study activities | 1
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Masimo SafetyNet Alert (MSNA)
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Feasibility of Masimo SafetyNet Alert (MSNA) in a Supportive Housing Program
Description: Number of participants who demonstrated feasibility of MSNA in a supportive housing program
Time Frame: 2-4 weeks
Population: 4 out of the 10 subjects were not completed due to physician decision, withdrawal by subject, or by death (unrelated to device, subject never participated in any study activities)
Measure: Number; unit: participants
Arm/Group | Masimo SafetyNet Alert (MSNA)
Number analyzed (Participants) | 10
participants | 6

2. Primary Outcome: Evaluation of Feasibility of Masimo SafetyNet Alert (MSNA) in a Supportive Housing Program
Description: Summarizing proportion of incomplete studies to evaluate the feasibility of Masimo SafetyNet Alert (MSNA) in a supportive housing program.
Time Frame: 2-4 weeks
Measure: Number; unit: incomplete studies
Arm/Group | Masimo SafetyNet Alert (MSNA)
Number analyzed (Participants) | 10
incomplete studies | 4

3. Primary Outcome: Evaluation of Feasibility of Masimo SafetyNet Alert (MSNA) in a Supportive Housing Program
Description: Summarizing proportion of lost components to evaluate the feasibility of Masimo SafetyNet Alert (MSNA) in a supportive housing program.
Time Frame: 2-4 weeks
Measure: Number; unit: lost components
Arm/Group | Masimo SafetyNet Alert (MSNA)
Number analyzed (Participants) | 6
lost components | 0

ADVERSE EVENTS:
Time Frame: Entirety of study (60 days)
Arm/Group | Masimo SafetyNet Alert (MSNA)
All-Cause Mortality (participants affected / at risk) | 1/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed. Some outcome measures could not be calculated due to small number of subjects being analyzed. No staff participants were enrolled in this study prior to termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2023-11-14): https://cdn.clinicaltrials.gov/large-docs/80/NCT06217380/Prot_001.pdf